CLINICAL TRIAL: NCT05545592
Title: A Randomized Controlled Trial on Reducing Oestrogen Dosage to Improve the Clinical Outcome of Frozen-thawed Embryo Transfer
Brief Title: Reduced Oestrogen Dosage to Improve the Outcome of Frozen-thawed Embryo Transfer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, principal investigator, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SZ-HRT-2022
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: FET

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low oestrogen (Experimental): The patients take orally estradiol tablets 2 mg (Femoston) q.d. during the HRT-FET cycles
  Interventions: Other: Low oestrogen dosage
- Regular oestrogen (No Intervention): The patients take orally estradiol tablets 2 mg (Femoston) t.i.d. during the HRT-FET cycles

INTERVENTIONS:
Other: Low oestrogen dosage — From the second day of the menstrual cycle, femoston (estradiol tablets) were orally taken 2 mg q.d.. The endometrial thickness and serum oestrogen and progesterone levels were monitored on the 12th to 14th days of the menstrual cycle.
  Arms: Low oestrogen

SUMMARY:
This study is a single-center, randomized, controlled prospective study. Those who will recieve hormone replacement therapy-frozen thawed embryo transfer (HRT-FET) are enrolled in the study. To determine the effect of oestrogen dosage reducion on maternal and fetal complications in HRT-FET cycles while maintaining the similar clinical pregnancy outcome in HRT-FET cycles with regular oestrogen dosage.

DETAILED DESCRIPTION:
According to the enrollment and exclusion criteria, the patients were enrolled, and the subjects were randomly divided into two groups by computer randomization. Group A was the reduced oestrogen dosage group (test group). Group B was the regular hormone replacement group (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Female;
2. Aged between 20 and 40 years old;
3. Frozen thawed embryo transfer is proposed, and the type of transferred embryo is blastocyst (the number of transferred embryos is 1);
4. Body mass index (BMI) ≤ 28 kg/m2, ≥ 18.5 kg/m2;
5. The total number of transfer cycles was < 3;
6. Volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Patients with chromosomal abnormalities;
2. Contraindications to hormone replacement therapy;
3. Patients with uterine myoma, severe adenomyosis, endometriosis, congenital uterine malformation, endometrial tuberculosis, intrauterine adhesions and other diseases that significantly affect embryo implantation;
4. Participating in other clinical studies.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 660 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 45 days after embryo transfer
  Clinical pregnancy is defined as the presence of gestational sac observed by ultrasound. The proportion of clinical pregnancy cycles to total FET cycles is the clinical pregnancy rate.

SECONDARY OUTCOMES:
Embryo implantation rate | 45 days after embryo transfer
  The proportion of the number of implanted embryos to the total number of transferred embryos is the embryo implantation rate.
Early pregnancy loss rate | 12 weeks after embryo transfer
  The early pregnancy loss rate refers to the proportion of patients with pregnancy loss before 12 weeks of gestation in the total clinical pregnancy patients.
Incidence of thrombosis | 12 weeks after embryo transfer
  Thrombosis incidence refers to the proportion of patients with deep venous thrombosis in the total patients.
Incidence rate of gestational hypertension | 45 weeks after embryo transfer
  The incidence rate of gestational hypertension refers to the proportion of patients with gestational hypertension in the total pregnant patients.
Premature birth rate | 41 weeks after embryo transfer
  Preterm birth rate refers to the proportion of patients with preterm birth in all pregnancies.
Proportion of low birth weight infants | 41 weeks after embryo transfer
  The proportion of low birth weight infants refers to the proportion of low birth weight infants in all newborns.

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Center, The affiliated Drum Towel Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China